CLINICAL TRIAL: NCT07354516
Title: A Masked, Randomized, Prospective Study of QLS-111-FDC in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Study of QLS-111-FDC in Open-Angle Glaucoma or Ocular Hypertension
Acronym: Firecrest
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QC-300
Record Dates: First submitted 2026-01-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: OAG - Open-Angle Glaucoma; OHT - Ocular Hypertension
Keywords: glaucoma; intraocular pressure (IOP); eye drops
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IP is packaged and labeled in a masked fashion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QLS-111-FDC ophthalmic solution (Experimental): QLS-111-FDC, PF FDC
  Interventions: Combination Product: QLS-111-FDC
- Latanoprost ophthalmic solution (Active Comparator): PF latanoprost 0.005%
  Interventions: Drug: Latanoprost (0.005%)

INTERVENTIONS:
Combination Product: QLS-111-FDC — QLS-111-FDC, a PF FDC administered by topical ophthalmic (TO) application for 14 days in the evening (QPM) in both eyes (OU).
  Arms: QLS-111-FDC ophthalmic solution
Drug: Latanoprost (0.005%) — PF latanoprost administered by TO application for 14 days QPM OU.
  Other Names: latanoprost ophthalmic solution 0.005%, PF
  Arms: Latanoprost ophthalmic solution

SUMMARY:
Firecrest study is evaluating the intraocular pressure (IOP)-lowering effect, safety, and tolerability of Qlaris' preservative free [PF], fixed-dose combination [FDC] investigational product (IP) in subjects with open-angle glaucoma (OAG) or ocular hypertension (OHT).

DETAILED DESCRIPTION:
14-day prospective, double-masked, active-controlled, randomized multicenter study comparing QLS-111-FDC and PF latanoprost. Study is comprised of 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* BCVA 1.0 logMAR or better in each eye (equivalent to 20/200)
* Diagnosis of mild to moderate OAG or OHT in at least one eye
* IOP ≥19 mmHg at 08:00 hour (H) at Qualification Visits following a run-in with PF latanoprost

Exclusion Criteria:

* History of active ocular disease other than mild to moderate OAG/OHT
* Prior use of any topical PGA without a clinically meaningful response
* Noncompliant with current ocular anti-hypertensive medications or unwilling to be compliant throughout the study
* Use of other topical ocular concomitant medications 30 days prior
* History of angle closure or a narrow angle, significant ocular trauma, ocular infection, uveitis, intraocular surgery in either eye.
* Central corneal thickness in either eye <470 or >630 μm
* Clinically significant systemic or psychiatric disease, chronic kidney disease, or hypertension, hypotension, or diabetes that is uncontrolled.
* Participation in any investigational study within 30 days prior to Screening
* Females who are pregnant, nursing, or not using birth control.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IOP | Over 15 days
  Change from baseline in IOP, lowering of IOP compared to baseline is desirable outcome.

SECONDARY OUTCOMES:
Ocular safety and tolerability | Over 15 days
  Incidence of ocular adverse events
Ocular comfort | Over 15 days
  Ocular comfort following study treatment as assessed by subject and using a visual analog scale (VAS) provided by the site at the treatment period visits. Subjects will grade their ocular comfort on a scale of 0 (extremely comfortable) to 100 (extremely uncomfortable) by placing a vertical mark on the horizontal line.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Wirostko, MD, Study Director — Qlaris Bio, Inc.

IPD SHARING:
Plan to Share IPD: No